CLINICAL TRIAL: NCT06253325
Title: An Observational Pilot Study for the Multi-Modality Risk Prediction and Early Identification of Critically Ill Septic Patients in the Emergency Department
Brief Title: Early Detection of At-risk Septic Patients
Acronym: MMICS
Status: Recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CRI0436
Record Dates: First submitted 2024-01-08; First posted 2024-02-12 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Twenty millilitres of whole blood will be collected. Plasma will be separated by centrifugation and stored at -80 degrees celsius until further analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients presenting to the Emergency Department with suspected sepsis: Patients who present with potential sepsis. This is characterised by their illness suspected to be from an infection and significantly unwell defined by one of two scoring systems, either the National Early Warning Score or quick Sequential Organ Failure Assessment
  Interventions: Diagnostic Test: Measuring tissue oxygenation; Diagnostic Test: Procalcitonin; Diagnostic Test: Mid-regional proadrenomedullin; Diagnostic Test: Hand-held video microscope

INTERVENTIONS:
Diagnostic Test: Measuring tissue oxygenation — Measuring oxygen content of arteries, capillaries and veins
Diagnostic Test: Procalcitonin — Blood test
  Other Names: PCT
Diagnostic Test: Mid-regional proadrenomedullin — Blood test looking at inflammation in the body
  Other Names: MR-proADM
Diagnostic Test: Hand-held video microscope — A handheld video microscope that looks at blood flow through the capillaries of the tongue

SUMMARY:
The purpose of this study is to determine whether additional investigations used in other parts of healthcare can be used in the Emergency Department to identify critically ill patients quicker than usual care.

DETAILED DESCRIPTION:
The investigators intend to recruit 56 patients with suspected sepsis who attend the Emergency Department. The investigators want to use a device to monitor tissue oxygen levels when they first come into the Emergency Department as well as the change in tissue oxygen levels when a tourniquet is applied for 3 minutes. The investigators will take novel blood tests when the patient is having their routine bloods. Finally, the investigators will use a special camera to take specialised pictures of the small blood vessels under the tongue which will show blood flow through these vessels. The investigators will follow the recruited patients and determine if our extra data is better at determining who needs critical care. A significant proportion of patients may be too unwell or too distressed to consent to be part of this study. At the earliest opportunity, the investigators will ask patients when they have been stabilised and are able to give consent. If they say no, they will be removed from the study and their care will not be affected by this decision.

The results could help us identify septic shock as early as possible so that these unwell patients are identified early and get the correct treatment they need. This could mean starting advanced treatments usually found in the Intensive Care Unit very early on in a patient's journey.

ELIGIBILITY:
Inclusion Criteria:

1. Differential diagnosis which includes infection
2. Change in the quick Sequential Organ Failure Assessment (qSOFA) ≥2 or National Early Warning Score 2 (NEWS2) score ≥5
3. Aged ≥18 years

Exclusion Criteria:

1. Traumatic injury
2. Rockwood frailty score ≥6
3. Critical care therapy previously believed to not be in patient's best interests
4. Critical care therapies-initiated pre-hospital. Critical care therapies defined as:

   4.1 Mechanical ventilation 4.2 Vasopressor/inotrope therapy 4.3 Sedation or a general anaesthetic 4.4 Pre-hospital transfusion of blood products 4.5 Extra-corporeal support
5. Advanced directive refusing critical care therapies.
6. Acute cardiac failure
7. Active gastrointestinal bleed
8. Massive pulmonary embolism
9. ICU admission declined by critical care team
10. Treated in an acute hospital <6 hours before presentation to the Emergency Department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to the Emergency Department with their illness possibly caused by sepsis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-08-06 (Estimated); Study Completion 2025-08-06 (Estimated)

PRIMARY OUTCOMES:
Differences in tissue oxygenation | Up to 4 hours (from baseline); 28 days (follow-up)
  The difference in tissue oxygen saturation (StO2) during the vascular occlusion test in the Emergency Department between septic patients who need critical care treatment (CCT) compared to patients requiring ward care. This will be measured in % change per second..

SECONDARY OUTCOMES:
Baseline of tissue oxygenation | Up to 4 hours (from baseline); 28 days (follow-up)
  The difference in tissue oxygen saturation (StO2) at baseline in the Emergency Department between septic patients who need critical care treatment (CCT) compared to patients requiring ward care. This will be measured in %.
Difference in blood flow of the micro-circulation (microvascular flow index) | Up to 4 hours (from baseline); 28 days (follow-up)
  Differences in the flow of blood through small blood vessels underneath the tongue between the difference between septic patients who need critical care treatment (CCT) compared to patients requiring ward care. This will be measured by the Microvascular Flow Index (arbitrary units) which is a validated measurement assessing micro-circulatory flow.
Difference in blood flow of the micro-circulation (perfused vessel density) | Up to 4 hours (from baseline); 28 days (follow-up)
  Differences in the flow of blood through small blood vessels underneath the tongue between the difference between septic patients who need critical care treatment (CCT) compared to patients requiring ward care. This will be measured by the perfused vessel density (measured in mm/mm2) which is a validated measurement assessing micro-circulatory flow.
Difference in blood lactate levels | Up to 4 hours (from baseline); 28 days (follow-up)
  The difference in the blood tests of lactate between septic patients who need critical care treatment (CCT) compared to patients requiring ward care
Difference in blood tests (MR-proADM) | Up to 4 hours (from baseline); 28 days (follow-up)
  The difference in the blood tests of MR-proADM between septic patients who need critical care treatment (CCT) compared to patients requiring ward care
Difference in blood tests (Procalcitonin) | Up to 4 hours (from baseline); 28 days (follow-up)
  The difference in the blood tests of Procalcitonin (PCT) between septic patients who need critical care treatment (CCT) compared to patients requiring ward care
Correlation of extra investigations with standard patient outcomes | Up to 4 hours (from baseline); 28 days (follow-up)
  Looking at whether tissue oxygenation, buccal microcirculation (blood flow under the tongue) and biomarkers and correlation with clinical outcomes such as organ failure (SOFA) scores, 28-day hospital mortality, and length of hospital and ICU stay.

CONTACTS AND LOCATIONS:
Overall Officials: Ahilanandan Dushianthan, PhD, Study Director — University Hospital Southampton NHS Foundation Trust; James N Ward, BM, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in a publication will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication

REFERENCES:
- [Background] Hernandez G, Ospina-Tascon GA, Damiani LP, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Granda-Luna V, Cavalcanti AB, Bakker J; The ANDROMEDA SHOCK Investigators and the Latin America Intensive Care Network (LIVEN); Hernandez G, Ospina-Tascon G, Petri Damiani L, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Cavalcanti AB, Bakker J, Hernandez G, Alegria L, Ferri G, Rodriguez N, Holger P, Soto N, Pozo M, Bakker J, Cook D, Vincent JL, Rhodes A, Kavanagh BP, Dellinger P, Rietdijk W, Carpio D, Pavez N, Henriquez E, Bravo S, Valenzuela ED, Vera M, Dreyse J, Oviedo V, Cid MA, Larroulet M, Petruska E, Sarabia C, Gallardo D, Sanchez JE, Gonzalez H, Arancibia JM, Munoz A, Ramirez G, Aravena F, Aquevedo A, Zambrano F, Bozinovic M, Valle F, Ramirez M, Rossel V, Munoz P, Ceballos C, Esveile C, Carmona C, Candia E, Mendoza D, Sanchez A, Ponce D, Ponce D, Lastra J, Nahuelpan B, Fasce F, Luengo C, Medel N, Cortes C, Campassi L, Rubatto P, Horna N, Furche M, Pendino JC, Bettini L, Lovesio C, Gonzalez MC, Rodruguez J, Canales H, Caminos F, Galletti C, Minoldo E, Aramburu MJ, Olmos D, Nin N, Tenzi J, Quiroga C, Lacuesta P, Gaudin A, Pais R, Silvestre A, Olivera G, Rieppi G, Berrutti D, Ochoa M, Cobos P, Vintimilla F, Ramirez V, Tobar M, Garcia F, Picoita F, Remache N, Granda V, Paredes F, Barzallo E, Garces P, Guerrero F, Salazar S, Torres G, Tana C, Calahorrano J, Solis F, Torres P, Herrera L, Ornes A, Perez V, Delgado G, Lopez A, Espinosa E, Moreira J, Salcedo B, Villacres I, Suing J, Lopez M, Gomez L, Toctaquiza G, Cadena Zapata M, Orazabal MA, Pardo Espejo R, Jimenez J, Calderon A, Paredes G, Barberan JL, Moya T, Atehortua H, Sabogal R, Ortiz G, Lara A, Sanchez F, Hernan Portilla A, Davila H, Mora JA, Calderon LE, Alvarez I, Escobar E, Bejarano A, Bustamante LA, Aldana JL. Effect of a Resuscitation Strategy Targeting Peripheral Perfusion Status vs Serum Lactate Levels on 28-Day Mortality Among Patients With Septic Shock: The ANDROMEDA-SHOCK Randomized Clinical Trial. JAMA. 2019 Feb 19;321(7):654-664. doi: 10.1001/jama.2019.0071. PMID 30772908
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Hylander Moller M, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock 2021. Crit Care Med. 2021 Nov 1;49(11):e1063-e1143. doi: 10.1097/CCM.0000000000005337. No abstract available. PMID 34605781
- [Background] Parrott F. Length of stay , survival and organ support of admissions with septic shock to adult , general critical care units in England , Wales and Northern Ireland. 2014.
- [Background] Liu Z, Meng Z, Li Y, Zhao J, Wu S, Gou S, Wu H. Prognostic accuracy of the serum lactate level, the SOFA score and the qSOFA score for mortality among adults with Sepsis. Scand J Trauma Resusc Emerg Med. 2019 Apr 30;27(1):51. doi: 10.1186/s13049-019-0609-3. PMID 31039813
- [Background] Sepsis: recognition, diagnosis and early management: (c) NICE (2017) Sepsis: recognition, diagnosis and early management. BJU Int. 2018 Apr;121(4):497-514. doi: 10.1111/bju.14179. No abstract available. PMID 29603898
- [Background] Jones S, Moulton C, Swift S, Molyneux P, Black S, Mason N, Oakley R, Mann C. Association between delays to patient admission from the emergency department and all-cause 30-day mortality. Emerg Med J. 2022 Mar;39(3):168-173. doi: 10.1136/emermed-2021-211572. Epub 2022 Jan 18. PMID 35042695
- [Background] Linder A, Arnold R, Boyd JH, Zindovic M, Zindovic I, Lange A, Paulsson M, Nyberg P, Russell JA, Pritchard D, Christensson B, Akesson P. Heparin-Binding Protein Measurement Improves the Prediction of Severe Infection With Organ Dysfunction in the Emergency Department. Crit Care Med. 2015 Nov;43(11):2378-86. doi: 10.1097/CCM.0000000000001265. PMID 26468696
- [Background] NHS Digital. Hospital Accident & Emergency Activity 2021-2022. 2022.
- [Background] Adhikari NK, Fowler RA, Bhagwanjee S, Rubenfeld GD. Critical care and the global burden of critical illness in adults. Lancet. 2010 Oct 16;376(9749):1339-46. doi: 10.1016/S0140-6736(10)60446-1. Epub 2010 Oct 11. PMID 20934212
- [Background] NHS England (NHS-E). Critical Care Bed Capacity and Urgent Operations Cancelled 2019-20 Data.
- [Background] Simpson HK, Clancy M, Goldfrad C, Rowan K. Admissions to intensive care units from emergency departments: a descriptive study. Emerg Med J. 2005 Jun;22(6):423-8. doi: 10.1136/emj.2003.005124. PMID 15911950
- [Background] Diagnostics Assessment Programme Diagnosis and monitoring of sepsis : procalcitonin testing ( ADVIA Centaur BRAHMS PCT assay , BRAHMS PCT Sensitive Kryptor assay , Elecsys BRAHMS PCT assay , LIAISON BRAHMS PCT assay. 2014.
- [Background] Dilken O, Ergin B, Ince C. Assessment of sublingual microcirculation in critically ill patients: consensus and debate. Ann Transl Med. 2020 Jun;8(12):793. doi: 10.21037/atm.2020.03.222. PMID 32647718
- [Background] Ait-Oufella H, Lemoinne S, Boelle PY, Galbois A, Baudel JL, Lemant J, Joffre J, Margetis D, Guidet B, Maury E, Offenstadt G. Mottling score predicts survival in septic shock. Intensive Care Med. 2011 May;37(5):801-7. doi: 10.1007/s00134-011-2163-y. Epub 2011 Mar 4. PMID 21373821
- [Background] Falotico JM, Shinozaki K, Saeki K, Becker LB. Advances in the Approaches Using Peripheral Perfusion for Monitoring Hemodynamic Status. Front Med (Lausanne). 2020 Dec 7;7:614326. doi: 10.3389/fmed.2020.614326. eCollection 2020. PMID 33365323
- [Background] Vorwerk C, Coats TJ. The prognostic value of tissue oxygen saturation in emergency department patients with severe sepsis or septic shock. Emerg Med J. 2012 Sep;29(9):699-703. doi: 10.1136/emermed-2011-200160. Epub 2011 Sep 21. PMID 21946179
- [Background] Haertel F, Reisberg D, Peters M, Nuding S, Schroeder J, Werdan K, Ebelt H. Prognostic Value of Tissue Oxygen Saturation Using a Vascular Occlusion Test in Patients in the Early Phase of Multiorgan Dysfunction Syndrome. Shock. 2019 Jun;51(6):706-712. doi: 10.1097/SHK.0000000000001225. PMID 30052575
- [Background] AnaesthesiaUK. Principles of pulse oximetry [Internet]. AnaesthesiaUK. 2004. Available from: https://www.frca.co.uk/article.aspx?articleid=332
- [Background] Lipcsey M, Eastwood GM, Woinarski NC, Bellomo R. Near-infrared spectroscopy of the thenar eminence: comparison of dynamic testing protocols. Crit Care Resusc. 2012 Jun;14(2):142-7. PMID 22697622
- [Background] Macdonald SP, Brown SG. Near-infrared spectroscopy in the assessment of suspected sepsis in the emergency department. Emerg Med J. 2015 May;32(5):404-8. doi: 10.1136/emermed-2013-202956. Epub 2013 Oct 23. PMID 24154943
- [Background] Pinsky MR. Functional hemodynamic monitoring. Crit Care Clin. 2015 Jan;31(1):89-111. doi: 10.1016/j.ccc.2014.08.005. PMID 25435480
- [Background] Guyette FX, Gomez H, Suffoletto B, Quintero J, Mesquida J, Kim HK, Hostler D, Puyana JC, Pinsky MR. Prehospital dynamic tissue oxygen saturation response predicts in-hospital lifesaving interventions in trauma patients. J Trauma Acute Care Surg. 2012 Apr;72(4):930-5. doi: 10.1097/TA.0b013e31823d0677. PMID 22491607
- [Background] De Backer D, Hollenberg S, Boerma C, Goedhart P, Buchele G, Ospina-Tascon G, Dobbe I, Ince C. How to evaluate the microcirculation: report of a round table conference. Crit Care. 2007;11(5):R101. doi: 10.1186/cc6118. PMID 17845716
- [Background] Thooft A, Favory R, Salgado DR, Taccone FS, Donadello K, De Backer D, Creteur J, Vincent JL. Effects of changes in arterial pressure on organ perfusion during septic shock. Crit Care. 2011;15(5):R222. doi: 10.1186/cc10462. Epub 2011 Sep 21. PMID 21936903
- [Background] Scorcella C, Damiani E, Domizi R, Pierantozzi S, Tondi S, Carsetti A, Ciucani S, Monaldi V, Rogani M, Marini B, Adrario E, Romano R, Ince C, Boerma EC, Donati A. MicroDAIMON study: Microcirculatory DAIly MONitoring in critically ill patients: a prospective observational study. Ann Intensive Care. 2018 May 15;8(1):64. doi: 10.1186/s13613-018-0411-9. PMID 29766322
- [Background] Massey MJ, Shapiro NI. A guide to human in vivo microcirculatory flow image analysis. Crit Care. 2016 Feb 10;20:35. doi: 10.1186/s13054-016-1213-9. PMID 26861691
- [Background] Andaluz-Ojeda D, Nguyen HB, Meunier-Beillard N, Cicuendez R, Quenot JP, Calvo D, Dargent A, Zarca E, Andres C, Nogales L, Eiros JM, Tamayo E, Gandia F, Bermejo-Martin JF, Charles PE. Superior accuracy of mid-regional proadrenomedullin for mortality prediction in sepsis with varying levels of illness severity. Ann Intensive Care. 2017 Dec;7(1):15. doi: 10.1186/s13613-017-0238-9. Epub 2017 Feb 10. PMID 28185230
- [Background] Saeed K, Legramante JM, Angeletti S, Curcio F, Miguens I, Poole S, Tascini C, Sozio E, Del Castillo JG. Mid-regional pro-adrenomedullin as a supplementary tool to clinical parameters in cases of suspicion of infection in the emergency department. Expert Rev Mol Diagn. 2021 Apr;21(4):397-404. doi: 10.1080/14737159.2021.1902312. Epub 2021 Mar 29. PMID 33736553
- [Background] Baldira J, Ruiz-Rodriguez JC, Wilson DC, Ruiz-Sanmartin A, Cortes A, Chiscano L, Ferrer-Costa R, Comas I, Larrosa N, Fabrega A, Gonzalez-Lopez JJ, Ferrer R. Biomarkers and clinical scores to aid the identification of disease severity and intensive care requirement following activation of an in-hospital sepsis code. Ann Intensive Care. 2020 Jan 15;10(1):7. doi: 10.1186/s13613-020-0625-5. PMID 31940096
- [Background] Ma H, Liu H, Wu C, Huang L. Diagnostic Value of Serum Heparin Binding Protein, Blood Lactic Acid Combined with hs-CRP in Sepsis and Its Relationship with Prognosis. Evid Based Complement Alternat Med. 2021 Nov 9;2021:5023733. doi: 10.1155/2021/5023733. eCollection 2021. PMID 34795784
- [Background] Royal College of Physicians. National Early Warning Score (NEWS) 2: Standardising the assessment of acute-illness severity in the NHS. Vol. 17, Updated report of a working party. London; 2017. 318-318 p.
- [Background] You JS, Park YS, Chung SP, Lee HS, Jeon S, Kim WY, Shin TG, Jo YH, Kang GH, Choi SH, Suh GJ, Ko BS, Han KS, Shin JH, Kong T; Korean Shock Society (KoSS) Investigators. Relationship between time of emergency department admission and adherence to the Surviving Sepsis Campaign bundle in patients with septic shock. Crit Care. 2022 Feb 11;26(1):43. doi: 10.1186/s13054-022-03899-0. PMID 35148797
- [Background] Massey MJ, Larochelle E, Najarro G, Karmacharla A, Arnold R, Trzeciak S, Angus DC, Shapiro NI. The microcirculation image quality score: development and preliminary evaluation of a proposed approach to grading quality of image acquisition for bedside videomicroscopy. J Crit Care. 2013 Dec;28(6):913-7. doi: 10.1016/j.jcrc.2013.06.015. Epub 2013 Aug 21. PMID 23972316